CLINICAL TRIAL: NCT02196129
Title: Immediate Pain Relieving Effects of Sinbaro-3 Pharmaco-acupuncture in Low Back Pain Patients; A Randomized Controlled Trial
Brief Title: Immediate Pain Relieving Effects of Sinbaro-3 for Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, Dr, Jaseng Hospital of Korean Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JS-CT-2014-02
Record Dates: First submitted 2014-07-11; First posted 2014-07-21 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Low Back Pain With Radiculopathy; Low Back Pain Without Radiculopathy; Herniated Intervertebral Disc
Keywords: low back pain; pharmacoacupuncture; sinbaro-3
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain | interventions — Harpagophytum extract LI 174

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sinbaro-3 (Experimental): 1cc Harpagophytum Procumbens(freeze drying) pharmacoacupuncture adminstered to 6 acupoints at the site of pain Administered once and once only before any interventions
  Interventions: Drug: Sinbaro-3
- Hwangryun(distillation) (Placebo Comparator): 1cc Hwangryun(distillation) pharmaco-acupuncture administered to 6 acupoints at the site of pain Administered once and once only before any other intervention
  Interventions: Drug: Hwangryun

INTERVENTIONS:
Drug: Sinbaro-3 — 1cc administered to site of pain(ashi acupoints), once and once only before any other intervention/if pain in both low back and extermities, the site of most pain
  Other Names: Harpagophytum Procumbens
  Arms: Sinbaro-3
Drug: Hwangryun — 1cc administered to site of pain(ashi acupoints), once and once only before any other intervention/if pain in both low back and extermities, the site of most pain
  Arms: Hwangryun(distillation)

SUMMARY:
The purpose of this study is to investigate the immediate pain relieving effects of sinbaro-3 pharmaco-acupuncture in patients with low back pain admitted for inpatient care

DETAILED DESCRIPTION:
60 patients with LBP with moderate to severe pain(NRS>6) were randomly allocated to 2 groups. The experimental group was treated with sinbaro-3 pharmacoacupuncture and the control group was treated with Hwangryun pharmacoacupuncture. All administrations were limited to 1 session, and comparisons of measurements were made before and after treatment. Primary outcomes were measured using the VAS scale. Post-treatment follow-up will be performed to measure primary outcomes at 30 minutes, 2hours, 4hours, and 6 hours after treatment. Before and after each measurement, the patients are asked to stand up and rotate their torso. At termination of the study, satisfaction levels of the patient's current status will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to a Korean Medicine hospital for low back pain with or without radiculopathy
* Age between 18 and 69
* NRS score of >6 on the day of the intervention
* Voluntary participation with written consent given to study consent form

Exclusion Criteria:

* Diagnosis of serious disease(s) which are possible causes of back pain such as malignancy, vertebral fracture, spinal infection, inflammatory spondylitis, cauda equina compression, etc.
* Prior diagnosis of other chronic disease(s) which could affect effectiveness or interpretation of treatment results such as cardiovascular disease, diabetic neuropathy, fibromyalgia, rheumatoid arthritis, Alzheimer's disease, epilepsy, etc.
* Progressive neurologic deficit(s) or concurrent severe neurological symptoms
* Unsuitable for or at risk of complications from acupuncture treatment such as patients with clotting disorders, severe diabetes with risk of infection, serious cardiovascular disease, or undergoing anticoagulant treatment, etc.
* Under prescription of corticosteroids, immuno-suppressant drugs, psychiatric medicine, or other medication considered unsuitable for subjects by the researcher
* Experience of gastroenteric complications after taking NSAIDs or currently undergoing treatment for digestive disorders
* During pregnancy or suspected pregnancy
* Subjects considered unsuitable for clinical trial by the researcher

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | At baseline
  The patient is asked to stand up and roatate the torso to the left and right, then asked to mark on the visual analogue scale the intensity of the pain they are experiencing
Visual Analogue Scale | 30 minutes following treatment
  The patient is asked to stand up and roatate the torso to the left and right, then asked to mark on the visual analogue scale the intensity of the pain they are experiencing
Visual Analogue Scale | 2 hours following treatment
  The patient is asked to stand up and roatate the torso to the left and right, then asked to mark on the visual analogue scale the intensity of the pain they are experiencing
Visual Analogue Scale | 4 hours following treatment
  The patient is asked to stand up and roatate the torso to the left and right, then asked to mark on the visual analogue scale the intensity of the pain they are experiencing
Visual Analogue Scale | 6 hours following treatment
  The patient is asked to stand up and roatate the torso to the left and right, then asked to mark on the visual analogue scale the intensity of the pain they are experiencing

SECONDARY OUTCOMES:
Satisfaction levels | 6hrs following treatment
  7-point Likert scale

OTHER OUTCOMES:
Expected treatment effects | At baseline
  The patients are asked to reply how effective they think the treatment is going to be on a 6-point Likert-scale

CONTACTS AND LOCATIONS:
Overall Officials: Joonshik Shin, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea